CLINICAL TRIAL: NCT06479902
Title: Effects of Core Stability Combined With Diaphragmatic Strengthening Exercises Among Asthmatic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FUI/CTR/2024/14
Record Dates: First submitted 2024-06-07; First posted 2024-06-28 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: Mild Intermittent Asthma

STUDY DESIGN:
Intervention Model Description: Quasi Interventional Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Core stabilization and Diaphragmatic Exercise Group (Experimental): The intervention consisted of 18 sessions over three weeks, following the FITT protocol. Each session included a warm-up (5 minutes), core stability exercises (15 minutes), diaphragmatic strengthening exercises (10 minutes), and cool-down (5 minutes), with rest intervals. Exercises progressed in difficulty on stable surfaces, tailored to each participant's tolerance. Warm-up exercises included activities like hopping and knee circles, while core stability exercises featured moves such as planks and side planks. Diaphragmatic exercises included diaphragmatic breathing in various positions.
  Interventions: Procedure: Core stability exercise; Procedure: Diaphragmatic Strengthening Exercise

INTERVENTIONS:
Procedure: Core stability exercise — Core stability exercises featured moves such as planks and side planks.
Procedure: Diaphragmatic Strengthening Exercise — . Diaphragmatic exercises included diaphragmatic breathing in various positions.

SUMMARY:
This is a quasi intervention study evaluating the effects of core stabilization exercises and diaphragmatic strengthening on thoracic kyphosis angle, diaphragmatic excursion, chest expansion, lung functioning (FEV1/FVC ratio) and quality of life, in individuals with mild intermittent or mild persistent asthma.

DETAILED DESCRIPTION:
This study evaluated the effects of core stabilization exercises and diaphragmatic strengthening on thoracic kyphosis angle, diaphragmatic excursion, chest expansion, lung functioning (FEV1/FVC ratio), and quality of life in individuals with mild intermittent or mild persistent asthma. Thirty-seven participants from Fauji Foundation Hospital Rawalpindi underwent assessments before and after an 18-session treatment regimen over three weeks. The measures included diaphragmatic excursion, thoracic kyphotic angle, chest expansion, spirometry, and asthma quality of life questionnaire. Statistical analysis was performed using SPSS version 21

ELIGIBILITY:
Inclusion Criteria:

* Age group: 18-34 years old
* Both males and females
* Individuals diagnosed with well controlled mild intermittent asthma or mild persistent asthma, at least six months prior based on referral from pulmonologist.
* Individuals who have weak core muscles
* Participating to the study in a voluntary basis

Exclusion Criteria:

* Level 3 and above asthmatics or status asthmaticus
* Any congenital deformities of chest wall
* Demonstrated neuromuscular or neurological deficit/disease of chest wall.
* Cardiopulmonary diseases including coronary artery disease, heart failure NYHA classification, valvular heart disease, cardiomyopathy, arrythmias, interstitial lung disease, COPD, pulmonary embolism, pulmonary hypertension, cancers, etc.
* Any recent cardiothoracic or abdominal surgery or sternotomy
* Recent history of the blunt chest wall or abdominal trauma
* Unstable hemodynamic parameters (arterial pressure >140mmhg systolic and >90mmhg for diastolic
* Pregnancy
* Previous or parallel participation in interventional programs
* Any psychiatric illnesses

Ages: 18 Years to 34 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2023-07-15 (Actual); Primary Completion 2024-04-18 (Actual); Study Completion 2024-05-24 (Actual)

PRIMARY OUTCOMES:
Thoracic Kyphosis Angle | 18 days
  Measured with Inclinometer
Diaphragmatic Excursion | 18 days
  Measured using Tape method
Chest Expansion | 18 days
  Measured using Tape method
FEV1/FVC ratio | 18 days
  Measured using Spirometer
Quality of Life of patient | 18 days
  Asthma Quality of Life Questionnaire with Standardized Activities. It is a 32-item Likert-type scale that measures the impact of asthma on daily activities, with scores ranging from 1 (severe impairment) to 7 (no impairment).

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation University College of Physical Therapy, Rawalpindi, Punjab Province, Pakistan